CLINICAL TRIAL: NCT06980649
Title: An Open-Label Biomarker Study of BHV-1300 in Graves' Disease
Brief Title: Study of BHV-1300 in Graves' Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHV1300-202
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Graves Disease
Keywords: Autoimmune thyroid disease; hyperthyroidism; anti thyroid drug; thyroid disease; autoimmune diseases; endocrine system diseases
MeSH Terms: conditions — Graves Disease; Hyperthyroidism; Thyroid Diseases; Autoimmune Diseases; Endocrine System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BHV-1300 (Experimental)
  Interventions: Drug: BHV-1300

INTERVENTIONS:
Drug: BHV-1300 — BHV-1300 is delivered subcutaneously (SC)

SUMMARY:
The purpose of this study is to determine if BHV-1300 is a safe treatment in participants with Graves' Disease and to explore its effect on disease-specific biomarkers.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants must have serologically confirmed Graves' Disease.

Key Exclusion Criteria:

1. History of hyperthyroidism not caused by Graves' Disease (e.g., toxic adenoma or toxic multinodular goiter) and/or history of thyroid storm within six weeks of the Baseline visit.
2. History of treatment with radioactive iodine or thyroid surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Serious AEs (SAEs), AEs leading to discontinuation, deaths | Baseline to Week 12
  To assess the safety and tolerability of BHV-1300. This objective will be measured by assessing the number of unique subjects with SAEs, AEs leading to discontinuation or deaths that are observed during the Open-label Treatment Phase (up to 12 weeks).
Number of participants with Grade 3-4 (CTCAE/DAIDS) treatment-emergent laboratory abnormalities | Baseline to Week 12
  To assess the safety and tolerability of BHV-1300. This objective will be measured by assessing the number of unique subjects with Grade 3 or 4 treatment-emergent laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (6):
  - Site-103, South Gate, California
  - Site-100, Miami, Florida
  - Site-104, Columbus, Georgia
  - Site-106, Houston, Texas
  - Site-101, Houston, Texas
  - Site-105, Shavano Park, Texas
- Australia (6):
  - Site-004, Fitzroy
  - Site-001, Kotara
  - Site-003, Melbourne
  - Site-008, Parkville
  - Site-006, St Leonards
  - Site-002, Torquay